CLINICAL TRIAL: NCT06703827
Title: Effects of the Online MCT Group on Persecutory Delusions and Cognitive Biases in Clients with First Episode of Psychosis.
Brief Title: Effects of Online Metacognitive Training Group on Distressing Beliefs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 323885
Record Dates: First submitted 2024-05-13; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-05

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: The proposed study is an experimental, multi-centre trial aiming to investigate the impact of online MCT group on participants' persecutory delusions and cognitive biases in Early Intervention for Psychosis Service in Kent. Participants will be allocated randomly to either MCT group or Treatment as Usual Group (TAU) and these two groups will be compared to each other. This study will use an online survey called Qualtrics (Qualtrics, Provo, UT) that will include quantitative measures that participants will be asked to complete.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The chief investigator will be responsible for administering baseline outcome measures but not facilitating the MCT group sessions to minimize the potential for bias. Consequently, the assessment after the intervention will be performed in a fully blind manner. Participants will be reminded not to reveal their group status to the post-intervention assessor in order to maintain the blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCT group (Experimental): Online MCT group (10 sessions) will be delivered by colleague CBT therapist (with previous experience of delivering MCT group) and assistant psychologist/clinical associate psychological practitioner, where all professionals will receive appropriate training by chief investigator. The group will also have one expert patient who attended the previous pilot group (at The NHS Trust) and is willing to help conduct the current MCT training. All psychology staff have experience in delivering psychological therapies and working with psychosis.
  The study will use qualitative data to refine the results of the quantitative findings by using follow-up semi-structured interviews to better understand the participants' experiences who had a minimum of 40% reduction of their persecutory delusions and/or cognitive biases and/or secondary measures (CHOICE and CORE-OM 34). The interviews will be conducted immediately post-intervention.
  Interventions: Behavioral: The metacognitive training group
- Treatment as Usual Group (TAU) (No Intervention): TAU group: Treatment as usual is the general treatment protocol for patients with first episode of psychosis in the Early Intervention in Psychosis Service, where most patients have antipsychotic medication and at least monthly contact with care coordinator, and at least 6 monthly outpatient appointment with a psychiatrist.

INTERVENTIONS:
Behavioral: The metacognitive training group — The MCT will consist of spending 90 minutes a week in a small online group setting working through a series of workshops. Participants will also be asked to complete homework each week and they will be supported with this. Interviews and questionnaires regarding symptoms and thinking errors will be used before and immediately after the intervention. The participants who attended the group and improved in their symptoms and thinking errors will be invited to an interview asking them what worked for them and how they found the group.
  Arms: MCT group

SUMMARY:
Psychosis is characterized by distorted perceptions of reality, often involving persecutory delusions. Research links these symptoms to cognitive biases like "jumping to conclusions." Despite mixed reviews of Cognitive Behavioral Therapy (CBTp) for psychosis, a study will explore metacognitive training (MCT) delivered online. This training will be tested over 10 weeks with participants from a psychosis service in Kent, assessing its effect through interviews and questionnaires before and after the program, focusing on symptom improvement and cognitive changes.

DETAILED DESCRIPTION:
Psychosis is described as disruptions to a person's beliefs and view of the world that make it challenging for them to establish what is a reality. Some people with psychosis experience persecutory delusions, which is a distressing belief that harm will happen to them by others.

Research indicated that certain errors in thinking (called cognitive biases, e.g.: jumping to conclusions) have been linked to psychotic symptoms in at high risk from psychosis. Studies reveal that certain errors in thinking may be causal factors for the development and maintenance of delusions.

National Institute of Health and Care Excellence recommends psychological interventions such as Cognitive Behavioural Therapy for a Psychosis (CBTp), but the efficacy of CBTp has been questioned, and small uptake by clients has also been discovered. This research is based on the metacognitive training delivered in groups, which is a psycho-educational programme targeting these thinking errors in psychosis. Research indicates that this training can be delivered online in a group to participants with psychosis, hence it offered a promising treatment approach in times of pandemic.

The participants will be recruited from an Early Intervention in Psychosis service in Kent and will take part in a ten week MCT or Treatment as Usual (TAU). The MCT will consist of spending 90 minutes a week in a small online group setting working through a series of workshops. Participants will also be asked to complete homework each week and they will be supported with this. Interviews and questionnaires regarding symptoms and thinking errors will be used before and immediately after the intervention. The participants who attended the group and improved in their symptoms and thinking errors will be invited to an interview asking them what worked for them and how they found the group.

ELIGIBILITY:
New inclusion criteria (after amendment):

* participants who have a diagnosis of a first episode of psychosis, schizophrenia spectrum, affective disorder with psychotic symptoms;
* all participants will need to score 3 or above on PANSS delusions (PANSS, Kay et al., 1987)
* are of age 18-65 years;
* are conversant in English and able to read in English;

New exclusion criteria (after amendment)

* current inpatient admission;
* below 18 years of age;
* moderate to severe learning disability;
* severe organic impairment;
* severe substance use disorder;
* inability to speak and write fluently in English (hindering their ability to complete standardized assessments and fully participate in the intervention).
* currently taking part in any other interventional research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2025-07-27 (Estimated); Study Completion 2025-09-27 (Estimated)

PRIMARY OUTCOMES:
The Psychotic Symptom Rating Scales (PSYRATS) created by Haddock et al. (1999) | 1 week pre intervention and 1 week post-intervention
  This scale to measures delusional beliefs and auditory hallucinations. The scale has demonstrated excellent inter-rater, test-retest reliability (Haddock et al 1999). Furthermore, its validity has been established through research on individuals experiencing a first episode of psychosis (Drake et al., 2007).
The Cognitive Biases Questionnaire for Psychosis (CBQp), developed by Peters et al. (2014) | 1 week pre-intervention and 1 week post-intervention
  It evaluates specific cognitive biases such as catastrophizing, dichotomous thinking, emotional reasoning, and jumping to conclusions by using thirty vignettes that depict everyday life scenarios. Participants are asked to rate the scenarios based on four response options. Peters et al. (2014) have determined that this questionnaire has good reliability and concurrent validity.
The Positive and Negative Syndrome Scale (PANSS) | 1 week pre-intervention and 1 week post-intervention
  This is demonstrated in various studies such as Moritz et al. (2011), Favrod et al. (2014), Moritz et al. (2013), and Briki et al. (2014). The PANSS is a 30-item interview assessment tool designed to evaluate the intensity of psychotic symptoms and has demonstrated high interrater reliability (Kay et al., 1987).
The Revised Green et al. Paranoid Thoughts Scale - 18 items (R-GPTS; Freeman et al., 2019) | 1 week pre-intervention and 1 week post-intervention
  It is an outcome measure that is used to assess the presence and severity of paranoid thoughts. It consists of 18 items and was revised by Freeman et al. in 2019. The R-GPTS is used to assess the severity of paranoid thoughts in individuals with a range of mental health conditions such as paranoia and schizophrenia. The results of the studies conducted by Freeman et al. (2019) provide evidence for the validity and reliability of the R-GPTS as a measure of paranoid thoughts. These findings suggest that the R-GPTS can be used with confidence in clinical and research settings to accurately assess the presence and severity of paranoid thoughts.
The Fast and Slow Thinking Questionnaire (FAST, Hardy et al., 2020) | 1 week pre-intervention and 1 week post-intervention
  It is a measure of reasoning biases in individuals with paranoid thoughts. The study by Hardy et al. (2020) showed that the FAST has good internal consistency and test-retest reliability. The FAST scores were significantly associated with other measures of paranoid thoughts and were able to differentiate between individuals with high and low levels of paranoia, demonstrating its concurrent and discriminant validity. These findings suggest that the FAST is a reliable and valid tool for assessing reasoning biases in individuals with paranoia.
Delusional conviction will be self-rated weekly post each MCT Module using a visual scale (adapted from Freeman et al.'s RCT, 2021) | 1 week pre-intervention, weekly questionnaires over 10 weeks after each intervention, and 1 week post-intervention
  Scale will ask respondents to state how strongly they believe their persecutory belief, ranging from 0 (no conviction in belief) to 100 conviction (total conviction in belief).
  Level of happiness will be self-rated weekly after each MCT Module using a visual scale that will ask respondents how happy they feel, ranging from 0 (not at all) to 100 (very much).

SECONDARY OUTCOMES:
The Clinical Outcomes in Routine Evaluation (CORE-OM 34; Evans et al., 2002) | 1 week pre-intervention and 1 week post-intervention
  It is a widely used measure of distress in the psychology department's Early Intervention for Psychosis Service, where the researcher will conduct the study. The highest possible score on the questionnaire is 136, which indicates extreme levels of distress. It has been established as a valid measure with robust outcomes (Evans et al., 2002).
The CHOICE short form measure (Greenwood et al., 2010) | 1 week pre-intervention and 1 week post-intervention
  It evaluates psychological recovery and has demonstrated strong psychometric properties. It is also regularly utilized in the local Trust and service. This questionnaire assesses changes within CBTp and may also be useful in measuring outcomes of MCT.

CONTACTS AND LOCATIONS:
Overall Officials: Kasia Wawrzyniak, Principal Investigator — City, University of London
Locations (1):
- Kent and Medway NHS and Social Care Partnership Trust, Maidstone, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD will only be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anticipated January 2025 till 30.09.2025
Access Criteria: Via University email, requests will be discussed with academic supervisor